CLINICAL TRIAL: NCT06765889
Title: Mindfulness-Based Intervention for Stress Reduction in Adult Singaporeans a Pilot Study
Acronym: MISRAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Human Development and Potential (IHDP), Singapore (Other)
Responsible Party: Principal Investigator, Alessandro Sparacio, Principal Investigator, Institute for Human Development and Potential (IHDP), Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-102
Record Dates: First submitted 2024-12-26; First posted 2025-01-09 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Mindfulness Meditation
Keywords: Mindfulness; Self-Administered Mindfulness; Mental Health; Stress; Decentralized Clinical Trial
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness intervention (Experimental): The mindfulness intervention will consist of three tracks of mindfulness practice adapted from a traditional Mindfulness-Based Stress Reduction (MBSR) protocol. The three mindfulness tracks will incorporate essential elements of mindfulness practice: a) cultivating attentional stability by directing focus to present-moment bodily experiences (Moore et al., 2012), and b) fostering mindful meta-awareness by nonreactively and nonjudgmentally observing and accepting experiences (Dahl et al., 2015).
  Interventions: Behavioral: Mindfulness intervention
- Sham meditation (Active Comparator): The sham meditation group will aim to be indistinguishable from meditation practice for newcomers (Zeidan et al., 2015). Non-specific elements of meditation, such as a soothing instructor's voice and terminology designed to create the expectation of authentic mindfulness meditation for those unfamiliar with the practice, will be emphasized.
  However, the instructions will deliberately exclude the training of the two fundamental cognitive/meta-cognitive processes crucial in mindfulness practice. This intentional omission will involve 1) removing any attentional stability by providing participants with no specific point to anchor their attention and 2) offering no guidance on cultivating mindful meta-cognitive qualities of attention. Participants in the mindfulness group will be taught to observe and accept their present-moment experience without judgment or reaction. In contrast, sham instructions will provide no such guidance.
  Interventions: Behavioral: Control condition

INTERVENTIONS:
Behavioral: Mindfulness intervention — The mindfulness intervention will consist of three tracks of mindfulness practice adapted from a traditional Mindfulness-Based Stress Reduction (MBSR) protocol. The three mindfulness tracks will incorporate essential elements of mindfulness practice: a) cultivating attentional stability by directing focus to present-moment bodily experiences (Moore et al., 2012), and b) fostering mindful meta-awareness by nonreactively and nonjudgmentally observing and accepting experiences (Dahl et al., 2015).
  Arms: Mindfulness intervention
Behavioral: Control condition — The sham meditation group will aim to be indistinguishable from meditation practice for newcomers (Zeidan et al., 2015). Non-specific elements of meditation, such as a soothing instructor's voice and terminology designed to create the expectation of authentic mindfulness meditation for those unfamiliar with the practice, will be emphasized. However, the instructions will deliberately exclude the training of the two fundamental cognitive/meta-cognitive processes crucial in mindfulness practice. This intentional omission will involve 1) removing any attentional stability by providing participants with no specific point to anchor their attention and 2) offering no guidance on cultivating mindful meta-cognitive qualities of attention. Participants in the mindfulness group will be taught to observe and accept their present-moment experience without judgment or reaction. In contrast, sham instructions will provide no such guidance.
  Arms: Sham meditation

SUMMARY:
This pilot study investigates self-administered mindfulness (SAM) as a stress reduction intervention, serving as a feasibility assessment for a larger multi-site trial. The research addresses gaps in mindfulness literature, particularly timely given that stress profoundly affects individuals' lives, shaping their thoughts, behaviors, and emotional experiences (Aldwin, 2007; Lazarus & Folkman, 1984), and plays a significant role in conditions like depression and anxiety (Yang et al., 2015).

The study implements a sham meditation control condition, improving upon passive controls that often yield inflated effect sizes (Patterson et al., 2016). The methodology incorporates both subjective measures, addressing limitations noted by Nichols et al. (2008), and heart rate variability (HRV) measurements. HRV has proven useful for its sensitivity to stress-induced changes (Goldberger et al., 2001), with higher values indicating better parasympathetic recovery (Shaffer & Ginsberg, 2017; Michels et al., 2013).

Set in Singapore, where stress management is a significant concern (Chodavadia et al., 2023), the study builds on Kabat-Zinn's (2003, 2006) definition of mindfulness. Unlike traditional programs, these interventions are more accessible (Spijkerman et al., 2016).

Recent meta-analyses show mixed findings: some identified small but significant effects (Cavanagh et al., 2018; Taylor et al., 2021), while others found no evidence of effectiveness after accounting for publication bias (Sparacio et al., 2024a). The study considers Singapore's unique cultural position (Li, Ngin, & Teo, 2007) and utilizes smartphone-based HRV monitoring, supported by research validating PPG technology (Guede-Fernández et al., 2020).

Through its comprehensive approach and robust design, this pilot study aims to establish a foundation for future research while providing insights into SAM's effectiveness as a stress reduction technique.

DETAILED DESCRIPTION:
This pilot study will implement a fully decentralized approach to investigate self-administered mindfulness (SAM) interventions, leveraging digital tools to streamline the research process without requiring physical interaction between research teams and participants. The decentralized framework particularly suits SAM interventions due to their inherent flexibility and seamless integration into participants' daily routines.

The study will address critical methodological gaps in mindfulness research through a rigorous randomized, double-blind, two-arm parallel-groups design. To differentiate between genuine effects and expectation-related processes, the study will employ a sham meditation control condition, where participants will be led to believe they are practicing meditation. This control condition will maintain structural equivalence with the mindfulness intervention while deliberately excluding two fundamental processes: attentional anchoring and guidance on cultivating mindful meta-cognitive qualities.

The study will utilize a comprehensive digital infrastructure for data collection and intervention delivery. The current clinical trial will be conducted over a three-day period and will be administered entirely remotely, with participants engaging from their homes by accessing a Qualtrics link.

For objective stress measurement, the study will utilize smartphone-based heart rate variability (HRV) assessment via a validated app employing photoplethysmogram (PPG) technology. This approach is consistent with established methods for assessing physiological markers of stress during resting states. The smartphone-based measurement strategy will enable participants to engage in the study from their homes, potentially enhancing ecological validity and participant retention.

The study will implement a robust system for participant management and data security. Phone numbers will be retained temporarily for specific operational purposes: preventing multiple submissions, facilitating study material delivery, and ensuring compensation via an electronic payment system. To maintain anonymity, all collected data except phone numbers will be de-identified. The study coordinator will implement checks for duplicate numbers to maintain data integrity.

Participants will be organized into cohorts of approximately 20 individuals, with recruitment continuing until the target sample size is reached. Each cohort will begin the study within three weeks of recruitment completion, ensuring efficient study progression while maintaining manageable group sizes for monitoring and support.

The mindfulness intervention will incorporate three distinct tracks adapted from traditional mindfulness protocols. These tracks will focus on two essential elements: cultivating attentional stability through present-moment bodily awareness and fostering mindful meta-awareness through nonreactivity and nonjudgmental observation. The selection of these components is based on established findings regarding effective stress regulation in mindfulness training.

The sham meditation control will be carefully designed to be indistinguishable from genuine meditation practice for newcomers, incorporating non-specific elements such as soothing voice and appropriate terminology. However, it will intentionally omit the core cognitive and meta-cognitive processes essential to mindfulness practice, providing neither specific attention anchoring nor guidance on mindful attention qualities.

The study will implement a comprehensive assessment protocol, including both psychological and physiological measures. Participants will complete assessments at consistent times between 9 AM and 9 PM daily. The protocol will include:

Baseline psychological assessments using validated instruments:

Neuroticism assessment Resilience measurement Mindfulness assessment, focusing on key facets of mindfulness based on recent confirmatory factor analysis

Daily pre- and post-intervention assessments:

Self-reported stress assessment Ecological Momentary Assessment (EMA) for real-time state evaluation HRV measurements using standardized protocols

End of study assessments:

Mindfulness assessment, focusing on key facets of mindfulness based on recent confirmatory factor analysis Perceived Awareness of Research Hypothesis (PARH) to control for demand characteristics Intervention credibility and expectancy evaluation Comprehensive feedback on protocol usability and participant experience Participants will receive detailed instructions for proper finger placement during HRV measurements. The app will automatically validate measurement quality, requiring repeat assessments (up to two additional attempts) if initial measurements fail quality standards. All HRV data will be saved in CSV format for subsequent analysis.

The decentralized approach aims to overcome traditional trial challenges such as geographical constraints, limited diversity, and logistical barriers that typically hinder participant engagement. This methodology will particularly benefit participants who may have difficulty accessing study locations or lack time to participate in traditional trials, potentially leading to a more diverse and representative study population.

This pilot investigation will serve as a feasibility assessment for a planned larger multi-site trial, with special attention paid to the credibility and usability of the survey-based methodology. Post-intervention questionnaires will collect participant feedback on survey instruction clarity, navigation ease, and overall user experience, informing methodology refinements for future larger-scale, fully decentralized studies on SAM.

Future Applications and Cultural Considerations Given Singapore's position at the intersection of Eastern and Western cultures, findings from this feasibility study will provide valuable insights for future international studies bridging diverse cultural contexts. The results will help establish a foundation for developing cost-effective, accessible stress management strategies while advancing our understanding of decentralized trial methodologies in mindfulness research.

The study's innovative approach to decentralized intervention delivery and data collection will provide valuable insights for future remote clinical trials, potentially influencing the design and implementation of similar studies across various behavioral interventions and cultural contexts.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 21 years old.
2. Possess a smartphone capable of running the study applications with internet access.
3. Be fluent in the English language.
4. Have sufficient vision and hearing to complete the study procedures.

Exclusion Criteria:

1. Engaged in meditation within the six months preceding the experiment.
2. Member of the research team or an immediate family member (defined as spouses, parents, children, or siblings, whether biological or legally adopted).
3. Currently taking psychoactive medications, including antidepressants, anxiolytics, hypnotics, or stimulants, or having used these medications in the past week.
4. History of major neurological or psychiatric disease within the past six months.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-02-11 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2025-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Sparacio, Principal Investigator — A*STAR IHDP
Locations (1):
- Brenner Centre for Molecular Medicine, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
All data collected in the research study will be de-identified. Electronic data will be stored on a secure, password-protected computer, accessible only to the researchers.
  Phone numbers collected for reimbursement purposes and to prevent re-attempts of the study will be deleted upon completion of data collection.
  De-identified research data will be stored and analyzed and may be used for future research and deposited in an online public repository.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the start of the project both hardcopy and electronic data will be retained for a maximum of 10 years, after which they will be destroyed. Any future research arising from the collected data will be subject to review by the relevant institutional review board.
Access Criteria: Access to research data will be restricted to the Principal Investigator (PI), and the study team. Access will be controlled and monitored through password-protected systems available only to authorized personnel.
URL: https://osf.io/7mnqd/

REFERENCES:
- [Derived] Sparacio A, Davies JN, Lee E, Schmitt JAJ. Feasibility and Acceptability of a Smartphone-Delivered Mindfulness Intervention for Stress Reduction in Adult Singaporeans: Pilot Randomized Controlled Trial. JMIR Ment Health. 2025 Aug 19;12:e77793. doi: 10.2196/77793. PMID 40828581

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindfulness Intervention | Sham Meditation
Started | 30 | 30
Completed | 29 (Only 1 participant discontinued after end of Day2 study procedures.) | 30
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Mindfulness Meditation: The intervention included three unique guided practices, each designed to strengthen attentional stability and meta-awareness-key mechanisms associated with effective mindfulness training and stress regulation (Moore et al., 2012; Dahl et al., 2015; Stein et al., 2020). The sessions focused on the following elements:
  Attentional Stability: Participants were guided to anchor their focus on present-moment bodily experiences, such as breath sensations, physical posture, or environmental stimuli, to enhance their ability to sustain attention without distraction.
  Mindful Meta-Awareness: The practice encouraged nonreactive and nonjudgmental observation of thoughts, emotions, and bodily sensations, fostering acceptance and self-regulation skills.
- Total: Total of all reporting groups
Arm/Group | Sham Meditation | Mindfulness Meditation | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.60 (12.20) | 36.20 (12.00) | 33.93 (12.18)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 12 | 26 | 38
  Female | 17 | 13 | 30
  Other | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 29 | 27 | 56
  Other | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Stress
Description: We will measure self-reported acute stress using the State-Trait Anxiety Inventory - Short Form (STAI-6), a validated 6-item version of the 40-item State-Trait Anxiety Inventory developed by Marteau and Bekker. The STAI-6 assesses current (state) anxiety symptoms using a 4-point Likert scale ranging from 1 (Not at all) to 4 (Very much). Example items include "I feel calm" and "I am tense." For data analysis, the mean score of the 6 items was calculated. Therefore, scores range from 1 to 4, with higher scores indicating greater levels of acute stress (worse outcome). In the table, the averaged score for STAI-6 at pre/post assessments for each of the three days of the intervention is provided. Results for the two conditions are provided.
Time Frame: Participants will complete the STAI-6 assessment six times throughout the trial, once per day on Days 1 through 3. On each day, they will report their STAI-6 levels twice: once before listening to the audio track and once immediately after listening
Population: We used a Bayesian latent growth curve model in **brms** to assess the effect of the mindfulness intervention on STAI-6 stress scores. The model included fixed effects for time (Pre vs. Post), condition (Mindfulness vs. Sham), their interaction, and Day as a covariate, with random slopes for time by participant. We applied weakly informative priors and used Bayes Factors (BF₁₀) to compare the full model to a null model, evaluating support for the intervention effect.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Mindfulness: The Mindfulness Intervention, using tracks recorded by a certified MBSR instructor, aimed to enhance attentional stability and meta-awareness. Over three days, participants engaged in practices designed to anchor their focus on the present moment. These included a formal body awareness meditation, an informal practice of mindfully brushing their teeth, and a breath awareness exercise. The core of this condition was nonjudgmental observation of one's thoughts, feelings, and bodily sensations.
- Sham: the Sham Meditation Condition was crafted to mimic the structure of the mindfulness intervention without its key therapeutic elements. The sham tracks actively discouraged attentional stability and meta-awareness. Instead of focusing on a single anchor, participants were encouraged to let their minds wander, engage in multitasking, and explore thoughts freely. The daily activities included associative thinking, brushing teeth while planning other tasks, and creatively expanding on a chosen thought.
Arm/Group | Mindfulness | Sham
Number analyzed (Participants) | 30 | 30
score on a scale
  Day 1 Pre | 1.89 (0.69) | 1.87 (0.75)
  Day1 Post | 1.59 (0.50) | 1.68 (0.58)
  Day 2 Pre | 1.96 (0.58) | 1.89 (0.76)
  Day 2 Post | 1.71 (0.57) | 1.69 (0.59)
  Day 3 Pre | 2 (0.57) | 1.91 (0.80)
  Day 3 Post | 1.63 (0.49) | 1.68 (0.61)
Statistical Analysis 1: Comparison: Mindfulness vs Sham; Test type: Other; Bayes Factor (BF₁₀) = 0.03

2. Secondary Outcome: Physiological Stress
Description: Heart Rate Variability. To assess parasympathetic activation, participants' heart rate variability (HRV) will be analyzed. HRV is widely recognized as a sensitive marker of stress, regulated by the autonomic nervous system in response to stressors (Goldberger et al., 2001). Participants will monitor their HRV using the 'Camera Heart Rate Variability' smartphone app, which employs Photoplethysmogram (PPG) technology. Notably, smartphone apps utilizing PPG for heart rate measurement have shown consistency with validated methods such as electrocardiography (ECG) in adult populations during resting states (Guede-Fernández et al., 2020) Participants will be instructed to place their index finger over the smartphone's camera and flash, ensuring both are fully covered. They will hold their finger in place for one minute to allow the device to record their heart rate variability (HRV).
Time Frame: Participants will assess their HRV values seven times over the course of the trial (from Day 1 to Day 3). The first measurement will be a test, the first and second measurement each day will be taken before and after listening to the audio track.
Reporting Status: Not Posted

3. Secondary Outcome: Ecological Momentary Assessment - (EMA)
Description: Participants will indicate their current state using a slider scale from 1 (not at all) to 100 (very much). The following questions will be used to assess various psychological and physical states:
  * "Right now, I feel mentally sharp" - to assess perceived cognitive ability.
  * "Right now, I feel fatigued" - to assess fatigue and exhaustion.
  * "Right now, I feel stressed" - to assess stress levels.
  * "Right now, I feel nervous" - to assess nervousness and tension.
  * "Right now, I feel depressed" - to assess depressive symptoms.
  * "Right now, I am in a good mood" - to assess positive affect and joy.
  * "I slept well last night" - to assess subjective sleep quality.
Time Frame: Participants will complete the Ecological Momentary Assessments (EMAs) six times throughout the trial, once per day on Days 1 through 3. On each day, they will report their EMAs levels twice: once before listening to the audio track and once immediately
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Usability of the Intervention
Description: To assess the usability and acceptability of the pilot trial, participants from both the mindfulness and sham conditions completed a questionnaire after the final session. It evaluated dimensions including ease of use, clarity, engagement, relevance, and willingness to continue use.
  Items were rated on a 5-point Likert scale (1 = Strongly Disagree to 5 = Strongly Agree), with higher scores indicating greater perceived usability.
Time Frame: One time, during day 3 of the clinical trial.
Population: We measure acceptability with means and SD for both groups as the intervention (except for the different audio) was equivalent across conditions (same app to measure HRV, same procedure etc).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Sham Meditation: The Sham Meditation Condition was crafted to mimic the structure of the mindfulness intervention without its key therapeutic elements. The sham tracks actively discouraged attentional stability and meta-awareness. Instead of focusing on a single anchor, participants were encouraged to let their minds wander, engage in multitasking, and explore thoughts freely. The daily activities included associative thinking, brushing teeth while planning other tasks, and creatively expanding on a chosen thought.
Arm/Group | Mindfulness | Sham Meditation
Number analyzed (Participants) | 30 | 30
score on a scale | 4.17 (0.55) | 4.17 (0.51)
Statistical Analysis 1: Comparison: Mindfulness; Test type: Other; Mean (of both conditions) = 4.17

5. Other Pre Specified Outcome: Perceived Awareness of the Research Hypothesis
Description: PARH; Rubin 2016 is a four-item quantitative self-report tool designed to assess the possible impact of demand characteristics in research settings. Its purpose is to assist in challenging the notion that observed effects can be attributed to demand characteristics. Participants provide their responses to these statements using a 7-point Likert-type scale, where the options range from strongly disagree (1) to strongly agree (7). Examples of statements include: "I was aware of the researchers' objectives in this study" and "I was uncertain about the researchers" intentions in conducting this research".
Time Frame: One time, during day 3 of the clinical trial.
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Credibility of the Intervention
Description: To evaluate credibility, participants responded to a two-part question: "If you were informed that you might have received either meditation training or control training, which type do you believe you received? (Meditation, Control)". Furthermore, we asked to participants how confident were about that answer on a scale from 0 to 10. In the following table we excluded answers where their confidence about the answer was <5
Time Frame: One time, during day 3 of the clinical trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness | Sham Meditation
Number analyzed (Participants) | 30 | 30
Participants
  Correct Group Identification | 18 | 6
  Wrong Group Identification | 10 | 11
  Excluded answers (confidence <5) | 2 | 13

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored/collected.
Groups:
- Both Conditions: No Adverse events were recorded.
Arm/Group | Both Conditions
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Several key limitations should be considered when interpreting these findings. First, while the sample size (n=60) was adequate for assessing feasibility, it was underpowered to detect subtle intervention effects or moderation by psychological traits. Second, generalizability is limited to English-speaking, predominantly Chinese Singaporean adults without mental health conditions, and results may not extend to other populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-26): https://cdn.clinicaltrials.gov/large-docs/89/NCT06765889/Prot_SAP_000.pdf